CLINICAL TRIAL: NCT05774808
Title: Fate of Moderate Secondary Mitral Regurgitation in Patients Undergoing Aortic Valve Surgery for Severe Aortic Regurgitation
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: MOSMIR-SAR
Record Dates: First submitted 2023-01-30; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Aortic Regurgitation; Functional Mitral Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement; Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aortic valve surgery only
  Interventions: Procedure: Aortic valve replacement
- Aortic valve + mitral valve surgery
  Interventions: Procedure: Aortic valve replacement; Procedure: Mitral valve annuloplasty

INTERVENTIONS:
Procedure: Aortic valve replacement — An aortic valve prosthesis is surgically implanted to treat AR
Procedure: Mitral valve annuloplasty — Surgical repair of the mitral valve in which a prosthetic ring is implanted to treat MR
  Groups: Aortic valve + mitral valve surgery

SUMMARY:
Patients with severe aortic regurgitation (AR) may be affected, in many cases, by a concomitant moderate or severe mitral regurgitation (MR). Tethering of the mitral valve leaflets and/or annular dilatation, both consequences of left ventricular dilatation, represent the most common mechanisms underlying the development of MR which can therefore be defined as "secondary" in this case.

When both mitral and aortic regurgitation are severe, patients show a decreased survival due to the pathophysiological consequences of the combination of these pathological conditions. In this case, surgery on both diseased valves is required to interrupt the natural history of the disease and is widely supported by current guidelines. On the other hand, little is known about the fate and prognostic implications of moderate MR secondary to severe AR and whether or not it should be treated at the time of aortic valve surgery. For this condition, the current guidelines do not provide specific recommendations, referring generically to the decision of the Heart Team.

To date, there are few data describing the evolution of moderate MR in patients undergoing surgery for severe AR and insufficient data to support recommendations regarding the treatment of moderate MR concurrently with treatment of AR, so that this decision is now entrusted to the evaluation of the Heart Team. It is therefore desirable to evaluate the outcomes of these patients.

The aim of this study is to evaluate the short- and long-term fate of secondary moderate MR in patients undergoing aortic valve replacement for severe AR.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Patients with severe aortic regurgitation (AR) AND moderate mitral regurgitation (MR).
* Patients underwent isolated aortic valve surgery (Study Group) or concomitant mitral valve surgery (Control Group) and
* Patients operated at the Cardiac Surgery Department of the San Raffaele Hospital from January 2004 to January 2019

Exclusion Criteria:

* Patient with more than moderate MR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by severe AR and moderate MR. The patients are divided in 2 groups: in the Study group, patients underwent isolated aortic valve surgery, while in the Control group, mitral valve surgery was also added.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Mortality for cardiac causes | Through study completion, an average of 7 years

SECONDARY OUTCOMES:
All causes mortality | Through study completion, an average of 7 years
Severe AR recurrency | Through study completion, an average of 7 years
Reintervention for severe AR recurrency | Through study completion, an average of 7 years
Reintervention for severe MR | Through study completion, an average of 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No